CLINICAL TRIAL: NCT00062283
Title: A Phase II, Open-Label, Non-Randomized, Multicenter, Single Agent Study of Intravenous SDX-102 for the Treatment of Patients With MTAP-Deficient Cancer
Brief Title: Alanosine in Treating Patients With Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: SALMEDIX-SDX-102-01; MSKCC-03029; CDR0000304677 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2009-12

CONDITIONS: Lung Cancer; Malignant Mesothelioma; Pancreatic Cancer; Sarcoma
Keywords: advanced malignant mesothelioma; recurrent malignant mesothelioma; metastatic osteosarcoma; recurrent osteosarcoma; recurrent adult soft tissue sarcoma; stage IV adult soft tissue sarcoma; chondrosarcoma; recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the pancreas; recurrent pancreatic cancer; stage III adult soft tissue sarcoma; stage II adult soft tissue sarcoma; stage IV pancreatic cancer
MeSH Terms: conditions — Lung Neoplasms; Mesothelioma, Malignant; Pancreatic Neoplasms; Sarcoma; Osteosarcoma; Chondrosarcoma; Carcinoma, Non-Small-Cell Lung | interventions — alanosine

INTERVENTIONS:
Drug: L-alanosine

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as alanosine use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase II trial is studying how well alanosine works in treating patients with soft tissue sarcoma, sarcoma of the bone, mesothelioma, non-small cell lung cancer, or pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rates in patients with methylthioadenosine phosphorylase (MTAP)-deficient cancer when treated with alanosine.
* Determine the time to response and duration of response in patients treated with this drug.
* Determine the progression-free survival of patients treated with this drug.
* Determine the pharmacodynamic activity of this drug in these patients, based on special imaging to measure tumor adenosine triphosphate depletion.
* Determine the pharmacokinetic activity of this drug in these patients.
* Determine the safety and tolerability of this drug in these patients.

OUTLINE: This is a nonrandomized, open-label, multicenter study.

Patients receive alanosine IV continuously on days 1-5. Treatment repeats every 21 days for up to 9 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed at 28 days.

PROJECTED ACCRUAL: A total of 50-145 patients (10-29 per tumor type) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed malignancy of any of the following types:

  * Soft-tissue sarcoma

    * High grade
    * Chemotherapy naïve or progressive or metastatic after no more than 2 prior cytotoxic treatment regimens (not including adjuvant therapy)
  * Sarcoma of the bone (including osteosarcoma* and chondrosarcoma)

    * High grade
    * Progressive or recurrent after no more than 2 prior cytotoxic treatment regimens
    * No newly diagnosed or chemotherapy naïve disease NOTE: *Prior treatment with cisplatin and doxorubicin required
  * Mesothelioma

    * Unresectable
    * Chemotherapy naïve or progressive after no more than 1 prior cytotoxic chemotherapy regimen
    * Not amenable to curative treatment with surgery

      * Evidence of gross unresectability includes, but is not limited to, direct extension into the chest wall, mediastinal or hilar lymphadenopathy, pulmonary or cardiac function that is inadequate to tolerate resection, and sarcomatoid or mixed histology
  * Non-small cell lung cancer

    * Stage III with malignant pleural or pericardial effusion, stage IV, or progressive after no more than 2 prior cytotoxic chemotherapy regimens
    * No newly diagnosed or chemotherapy naïve disease
  * Pancreatic cancer

    * Stage IV adenocarcinoma after no more than 1 prior cytotoxic treatment regimen
    * No newly diagnosed or chemotherapy naïve disease
* No Ewing's sarcoma of the soft tissue or bone
* Documented absence of methylthioadenosine phosphorylase on fixed tumor specimens
* Measurable disease

  * For all tumor types, at least 1 lesion measurable by MRI or CT scan
  * Chest x-ray allowed only for clearly defined lesions surrounded by aerated lung
  * Soft tissue component of bone disease considered measurable provided it can be measured by MRI or CT scan
  * Must be outside of a previously irradiated area
* No uncontrolled CNS metastases of primary tumor under study

  * Patients with brain metastases are eligible only if the brain metastases have been treated with prior radiotherapy and/or surgery, are neurologically stable with no progressing symptoms, and are off steroids and anticonvulsants

PATIENT CHARACTERISTICS:

Age

* 18 and over (13 and over for osteosarcoma only)

Performance status

* WHO 0-2

Life expectancy

* At least 3 months

Hematopoietic

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2.5 times ULN
* AST and ALT no greater than 2.5 times ULN (5 times ULN if liver metastases are present)

Renal

* Creatinine no greater than 1.5 times ULN

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 4 weeks after study treatment
* No premalignant bony lesions (e.g., Paget's disease)
* No other concurrent active malignancy except completely excised nonmelanoma skin cancer or carcinoma in situ of the cervix or bladder
* No serious infection
* No medical or psychiatric condition that would preclude the achievement of the study objectives

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* More than 42 days since prior nitrosoureas or mitomycin

Endocrine therapy

* See Disease Characteristics

Radiotherapy

* See Disease Characteristics
* At least 28 days since prior brain radiotherapy
* More than 28 days since prior radiotherapy to more than 50% of the bone marrow

Surgery

* See Disease Characteristics
* At least 28 days since prior thoracic or other major surgery

Other

* Recovered from prior therapy
* More than 28 days since prior cytotoxic agents
* More than 28 days since prior anticancer investigational agents
* No other concurrent anti-tumor treatment

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-03; Primary Completion 2005-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul A. Meyers, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (12):
- United States (12):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Wilshire Oncology Medical Group, Incorporated - La Verne, La Verne, California
  - Cedars-Sinai Comprehensive Cancer Center at Cedars-Sinai Medical Center, Los Angeles, California
  - Lynn Regional Cancer Center West, Boca Raton, Florida
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Midwest Cancer Research Group, Incorporated, Skokie, Illinois
  - St. Vincent's Comprehensive Cancer Center - Manhattan, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Vanderbilt-Ingram Cancer Center at Vanderbilt Medical Center, Nashville, Tennessee
  - MD Anderson Cancer Center at University of Texas, Houston, Texas
  - U.S. Oncology, Incorporated, Houston, Texas